CLINICAL TRIAL: NCT03574441
Title: Intrapartum Epidural Catheter Displacement: Comparison of Three Dressing Methods in Morbidly Obese Parturients
Brief Title: Intrapartum Epidural Catheter Displacement: Dressing Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor Department of Anesthesiology and Perioperative Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1048027
Record Dates: First submitted 2018-06-01; First posted 2018-07-02 (Actual); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Analgesia, Obstetrical
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Patients were randomized using a random number table to be allocated to one of three groups with sealed envelopes, based on the type of dressing to be used to secure the epidural catheter after its insertion:
  1. TegadermTM plus catheter support pad.
  2. Dressing with TegadermTM plus Steri-StripTM bands
  3. Dressing with TegadermTM only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- TegadermTM only (Active Comparator)
  Interventions: Device: Tegaderm dressing only
- Dressing with TegadermTM plus Steri-StripTM bands (Active Comparator)
  Interventions: Device: Tegaderm dressing + Steri-strip dressing
- Dressing with TegadermTM plus catheter support pad. (Experimental)
  Interventions: Device: Tegaderm dressing + catheter support pad

INTERVENTIONS:
Device: Tegaderm dressing + catheter support pad — Tegaderm TM is a transparent tape. This intervention adds a support pad that comes in the epidural kit to help secure the catheter
  Arms: Dressing with TegadermTM plus catheter support pad.
Device: Tegaderm dressing + Steri-strip dressing — Tegaderm TM is a transparent tape. This intervention adds Steri Strips TM of tape to help secure the catheter
  Arms: Dressing with TegadermTM plus Steri-StripTM bands
Device: Tegaderm dressing only — Tegaderm TM is a transparent tape. This intervention uses only Tegaderm to secure the catheter
  Arms: TegadermTM only

SUMMARY:
Failure of labor epidural is a well-recognized situation in obstetric anesthesia practice. Incidence of epidural failure was shown to be 12% in a retrospective analysis of 19,259 deliveries. Epidural migration has been documented in both the obstetric and non-obstetric settings. It has been argued that prevention of epidural displacement is a potential remedy to at least part of the incomplete or failed epidurals in obstetrics.

Purpose: The investigators propose this study to prospectively evaluate the efficacy of the three types of epidural catheter dressings that are currently in use in clinical practice, in terms of catheter migration, taking into consideration the influence of body mass index on this variable.

DETAILED DESCRIPTION:
Primary aim: The investigators will evaluate the efficacy of three different epidural catheter dressing systems in laboring patients.

Secondary aims: To compare the effect of different degrees of obesity measured by BMI, on epidural catheter migration and quality and failure of epidural labor analgesia. To evaluate the effect of time an indwelling catheter remains in place, level of insertion and patient's height on epidural catheter migration.

Hypothesis: The use of dressing with transparent TegadermTM plus catheter support pad dressing is superior to the dressing with TegadermTM plus Steri-StripTM bands, and to a dressing with TegadermTM only, for epidural catheter fixation in laboring obese and morbidly obese patients, in terms of catheter migration. epidural quality and failure and epidural catheter replacement in the labor analgesia setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the Labor and delivery Unit at Augusta University Medical Center who request epidural analgesia.
2. BMI >30 kg/m2.
3. Age older than 18 years old.

Exclusion Criteria:

1. Allergy to adhesive tape or to the components of the dressings used in the study.
2. Preexisting sensory neurologic deficits affecting lower extremities.
3. Patients taken to the operating room for cesarean section during the study period.
4. Chronic pain conditions.
5. Patients with intrathecal catheters.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female
Enrollment: 91 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TegadermTM Only | Dressing With TegadermTM Plus Steri-StripTM Bands | Dressing With TegadermTM Plus Catheter Support Pad.
Started | 31 | 30 | 30
Completed | 31 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TegadermTM Only | Dressing With TegadermTM Plus Steri-StripTM Bands | Dressing With TegadermTM Plus Catheter Support Pad. | Total
Number analyzed (Participants) | 31 | 30 | 30 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 30 | 91
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 33] | 24 [18 to 32] | 25 [18 to 35] | 24 [18 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 30 | 91
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 19 | 20 | 61
  White | 9 | 11 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 30 | 91
Gestational age [Mean (Full Range); unit: Weeks] | 36 [33 to 39] | 37 [34 to 39] | 37 [34 to 40] | 36 [33 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Epidural Catheter Migration
Description: Percentage of participants for whom catheter migration was observed
Time Frame: 24 hours. The time from insertion to removal of catheter
Measure: Number; unit: percentage patients catheter migration
Arm/Group | TegadermTM Only | Dressing With TegadermTM Plus Steri-StripTM Bands | Dressing With TegadermTM Plus Catheter Support Pad.
Number analyzed (Participants) | 31 | 30 | 30
percentage patients catheter migration | 44 | 25 | 17

2. Secondary Outcome: Rate of Epidural Catheter Replacement
Description: Frequency of epidural catheter replacement due to analgesic failure among the catheters in each arm
Time Frame: 24 hours. The time from insertion to removal of catheter due to failure
Measure: Number; unit: percentage of catheters
Arm/Group | TegadermTM Only | Dressing With TegadermTM Plus Steri-StripTM Bands | Dressing With TegadermTM Plus Catheter Support Pad.
Number analyzed (Participants) | 31 | 30 | 30
percentage of catheters | 3.2 | 3.3 | 3.3

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | TegadermTM Only | Dressing With TegadermTM Plus Steri-StripTM Bands | Dressing With TegadermTM Plus Catheter Support Pad.
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03574441/Prot_SAP_000.pdf